CLINICAL TRIAL: NCT06383182
Title: Change in Serum Biomarkers After Endovascular Treatment for Acute Anterior Circulation Large Vessel Occlusion: a Prospective, Registry Study
Brief Title: Change in Serum Biomarkers After Endovascular Treatment for Acute Anterior Circulation Large Vessel Occlusion
Status: Recruiting | Type: Observational
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Director, General Hospital of Shenyang Military Region
Other Study IDs: Y (2024) 054
Record Dates: First submitted 2024-04-17; First posted 2024-04-25 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: endovascular treatment — all patients with anterior circulation large vessel occlusion will receive endovascular treatment.

SUMMARY:
Acute ischaemic stroke (AIS) results in high rates of neurological morbidity and mortality, especially in patients with large vessel occlusion (LVO). Endovascular therapy (EVT) has been approved as the most effective treatment for patients with LVO , but about half patients undergoing EVT did not achieve good outcome. The mechanisms of poor prognosis are complex. How to accurately identify serological biomarkers related to patients' clinical prognosis is an important research topic nowadays.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-80 years;
2. Patients with acute anterior circulation large vessel occlusion within 24 hours of onset who will receive endovascular treatment;
3. Pre-stroke mRS: 0-1;
4. Baseline NIHSS: ≥6;
5. Signed informed consent.

Exclusion Criteria:

1. The presence of contraindications to internal jugular vein cannulation;
2. Receiving intravenous thrombolysis;
3. Haemorrhagic stroke (cerebral haemorrhage or subarachnoid haemorrhage);
4. Coagulation disorders, systemic bleeding tendency, thrombocytopenia (<100×109/L);
5. Severe cardiac, hepatic or renal insufficiency (ALT or AST elevated more than 2 times the upper limit of normal value, or serum creatinine elevated more than 1.5 times the upper limit of normal value or in need of dialysis) or other serious medical diseases;
6. Severe uncontrolled hypertension (systolic blood pressure greater than 200 mmHg or diastolic blood pressure greater than 110 mmHg);
7. Pregnant or lactating women;
8. Other conditions who are not suitable for this trial by investigator.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with acute anterior circulation large vessel occlusion within 24 hours of onset who will receive endovascular treatment
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-07-02 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Dynamic changes in serum biomarkers after endovascular treatment | from the baseline to immediately, 30 minutes, 6 hours, and 24 hours after endovascular treatment
  These biomarkers will be identified based on proteomic methods

SECONDARY OUTCOMES:
favourable functional outcome, defined as modified Rankin Scale (mRS) 0-2 | 90±7 days
  mRS ranges from 0-6, high score means poor outcome
excellent functional outcome, defined as modified Rankin Scale (mRS) 0-1 | 90±7 days
  mRS ranges from 0-6, high score means poor outcome
distribution of modified Rankin Scale (mRS) score | 90±7 days
  mRS ranges from 0-6, high score means poor outcome
early neurological improvement, defined as 4 or more decrease in National Institute of Health stroke scale (NIHSS) | 24±8 hours
  NIHSS ranges from 0-22, with high score meaning severe neurological deficit.
changes in National Institute of Health stroke scale (NIHSS) | 24±8 hours
  NIHSS ranges from 0-22, with high score meaning severe neurological deficit.
symptomatic intracranial hemorrhage (sICH) | 24±8 hours
  sICH is defined as an increase in 4 or more points on the NIHSS
occurence of new stroke or other vascular events | 90±7 days

OTHER OUTCOMES:
the association between cerebral circulation time (CCT) and clinical outcomes | 24±8 hours, 10±2 days, 90±7 days
  CCT is defined as the time from the appearance of contrast at the siphon segment of the internal carotid to the end of the arterial phase during DSA on the anteroposterior and lateral image in anterior circulation LVO; clinical outcomes include changes in NIHSS and mRS
the association between serum biomarkers and clinical outcomes | 24±8 hours, 10±2 days, 90±7 days
  serum biomarkers include those in different timepoints or their dynamic changes; clinical outcomes include changes in NIHSS and mRS
the association between serum biomarkers and status of vessel recanalization | 24±8 hours, 10±2 days, 90±7 days
  serum biomarkers include those in different timepoints or their dynamic changes; the status of vessel recanalization is determined by modified thrombolysis in cerebral infarction

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Northern Theater Command, Shenyang, China

IPD SHARING:
Plan to Share IPD: Undecided